CLINICAL TRIAL: NCT06044363
Title: Assessing the Efficacy and Acceptability of the Satir Model on Self-esteem and Mental Health Among Individuals With Substance Use Disorders in China: A Pilot Study Protocol
Brief Title: Satir Model for Self-esteem, Mental Health, and Family Function Among Individuals With Substance Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Polly MA Haixia, Assistant Professor, Hong Kong Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HE-SF2023/26
Record Dates: First submitted 2023-09-11; First posted 2023-09-21 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Drug Abuse; Self Esteem; Mental Health Wellness 1; Family Dysfunction
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: a single center, open-label, randomized, controlled trial
Who Masked: Participant
Masking Description: Open trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Satir group (Experimental): Participants in the intervention group will receive a 10-session Satir model intervention.
  Interventions: Other: Satir group
- Control group (No Intervention): Participants in the control group will receive care as usual.

INTERVENTIONS:
Other: Satir group — Participants in the intervention group will receive a 10-session, 3-hour/session intervention that spans over a period of five days (2 sessions/day). The intervention program will be conducted on specific weekends, with a gap of 1 to 2 weeks. The total duration of the intervention will be 30 hours.
  Arms: Satir group

SUMMARY:
Self-esteem and family functioning are associated with mental health and success of drug treatment among individuals with substance use disorders (SUD). The Satir model aims to empower individuals to explore their internal resources, address emotional issues, shift coping strategies, enhancing self-esteem, and develop healthier ways of relating to themselves and others. It offers a range of techniques to enhance self-esteem, challenging negative belief systems, and promote personal growth. The aim of the study is to investigate the acceptability and preliminary efficacy of the Satir model on self-esteem, mental health, and family function among individuals with SUD in China. The study will adopt a mixed-method approach. The quantitative phase will employ a randomized control trial (RCT) utilizing a pre-post study design. The qualitative phase will involve conducting semi-structured individual interviews.The data will be analyzed by using SPSS software package (IBM SPSS statistics version 26.0). The individual-interview will be analyzed by using the six-phase thematic analysis. The study has the potential to advance knowledge in the field of drug rehabilitation interventions, inform evidence-based practice, and improve the wellbeing and outcomes of individual with SUD. It can contribute to the ongoing efforts to address the complex challenges associated with substance use and support individual on their trajectory to recovery.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 or above;
2. are able to speak, read, and write Chinese;
3. are willing to participate in the study and share their experience of the intervention with the research group;
4. have informed consent to participate in the study.

Exclusion Criteria:

1. have been diagnosed with severe mental illnesses, such as schizophrenia, mania, antisocial personality disorder;
2. have a diagnosed memory and cognitive impairment;
3. are undergoing psychotherapeutic or psychopharmacologic treatment;
4. are participating in similar studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-09-09 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Self-esteem | Through study completion, an average of two months
  The changes of participants' self-esteem will be assessed by using the Chinese version of Rosenberg self-esteem scale. Total scores range from 10 to 40, with higher scores representing lower self-esteem.

SECONDARY OUTCOMES:
Adult attachment | Through study completion, an average of two months
  Adult attachment will be assessed by using Adult attachment scale (AAS).The scale consists of 18 items scored on a 5 point likert-type scale. It measures adult attachment styles named "Secure", "Anxious" and "Avoidant".
Coping style | Through study completion, an average of two months
  Coping style via Chinese version of simplified coping style questionnaire (SCSQ). It consists of 20 items referring to different ways of coping, with a total score range from 0 to 60. Two subscales are active coping and passive coping.
Self-efficacy | Through study completion, an average of two months
  self-efficacy will be assessed by the general self-efficacy scale (GSES). The total score range from 10 to 40. Higher scores indicate higher perceived general self-efficacy
Meaning in life | Through study completion, an average of two months
  Meaning in life will be assessed by using the Chinese version of meaning in life questionnaire (MLQ). It includes 10 items with a total score range from 10 to 70. It consists two subscales: MLQ Presence (MLQ-P) and Search (MLQ-S), each of them containing five items. The internal consistency of MLQ is 0.819.
Resilience | Through study completion, an average of two months
  Resilience will be assessed via. the 25-item Connor-Davidson Resilience Scale (CD-RISC-25). The items are evaluated on a five-point likert scale ranging from 1 to 4. These ratings result in a number between 0-100, and higher scores indicate higher resilience.
Positive and negative affect scale | Through study completion, an average of two months
  Positive and negative affect scale via Positive and negative affect scale (PANAS). This brief scale is comprised of 20 items, with 10 items measuring positive affect (e.g., excited, inspired) and 10 items measuring negative affect (e.g., upset, afraid). Scores can range from 10 to 50 for both the Positive and Negative Affect, with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect.
Drug craving | Through study completion, an average of two months
  Drug craving will be assessed via the drug craving scale. It measures five dimensions of substance craving, including (1) prizing substance craving; (2) reflecting substance craving; (3) social substance craving; (4) negative substance craving; and (5) eliminating substance craving. The items are evaluated on a seven-point likert scale ranging from 1(strongly disagree) to 7 (strongly agree),
Motivation to abstain from drugs | Through study completion, an average of two months
  Motivation to abstain from drugs will be assessed via the motivation to abstain from drugs. It includes 31 items, The items are evaluated on a five-point likert scale ranging from 1(strongly disagree) to 5 (strongly agree), with higher score indicates higher level of motivation to abstain from drugs.
Family function | Through study completion, an average of two months
  Family function via the Chinese version of the 60-item McMaster Family Assessment Device (FAD). It includes seven subscale: problem solving, communication, roles, affective responsiveness, affective involvement, behavior control, and general function. The higher the overall score, the worse the level of family function.

CONTACTS AND LOCATIONS:
Overall Officials: Haixia Ma, PhD, Principal Investigator — Hong Kong Metropolitan University
Locations (1):
- Fangqiang compulsory isolation detoxification center, Yancheng, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized participant-level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Supporting Information: SAP, ICF, CSR
Time Frame: After the project is completed and the results of the project have been published.
Access Criteria: Request could be sent to Principal Investigator (phxma@hkmu.edu.hk)